CLINICAL TRIAL: NCT06870370
Title: Role of Non-Selective Beta-Adrenergic Blocker in Severe Traumatic Brain Injury
Brief Title: Role of Non-Selective Beta-Adrenergic Blocker in Severe TBI
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Huda Talaat Ibrahim Elkallaf, Resident of Emergency Medicine and Traumatology, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 36264MS291/8/23
Record Dates: First submitted 2025-03-06; First posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Traumatic Brain Injury (TBI) Patients; Intracranial Pressure; Intensive Care Unit; Mortality
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Propranolol; Control Groups

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Propranolol group (Experimental): This group Will receive propranolol intravenously at a dose of 1 mg every 6 h for 7 days.
  Interventions: Drug: propranolol
- normal saline IV group (Placebo Comparator): This group Will receive 1ml of sterile 0.9% normal saline IV every 6 hours for 7 days
  Interventions: Drug: normal saline IV

INTERVENTIONS:
Drug: propranolol — This group Will receive propranolol intravenously at a dose of 1 mg every 6 h for 7 days, and doses will be held if heart rate less than 60 bpm, mean arterial pressure less than 65 mmHg
  Other Names: Experimental group
  Arms: Propranolol group
Drug: normal saline IV — This group Will receive 1ml of sterile 0.9% normal saline IV every 6 hours for 7 days
  Other Names: control group
  Arms: normal saline IV group

SUMMARY:
The role of nonselective beta adrenergic blocker as antistress agent in severe traumatic brain injury

DETAILED DESCRIPTION:
The primary injury occurs at the time of trauma. secondary injury is caused by complications of the primary insult and caused by processes such as hypoxia, cerebral edema and ischemia.

Severe traumatic brain injury is associated with increased intracranial pressure, activation of the sympathetic nervous system and catecholamine response and major morbidity and mortality .

β-blockade is just one pharmacologic strategy to reduce sympathetic hyperactivity. In the Intensive care unit patients with severe traumatic brain injury associated with restlessness and agitation are frequently sedated and intubated in order to reduce the workload of the brain. This hyperactive response is called sympathetic storming which occurs within 24 hours of brain injury or weeks later . It occurs due to acceleration in sympathetic nervous system activity in the central nervous system which results in loss of cortical control due to downregulation of autonomic balance in the brain injury .

A Non-Selective beta-adrenergic antagonist propranolol, is one of the most customarily used treatments in the case of paroxysmal sympathetic hyperactivity.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18and 65 years old
* Patients who have Severe traumatic brain injury
* Glascow outcome scale ≤ 8

Exclusion Criteria:

* Patients have pre-existing heart disease.
* If there are contraindications to β blocker.
* penetrating traumatic brain injury.
* pre-injury brain dysfunction.
* β-blocker or α2-agonist use before trauma.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-09-20 (Estimated); Primary Completion 2025-09-20 (Estimated); Study Completion 2025-09-20 (Estimated)

PRIMARY OUTCOMES:
Mortality | 7 days
  Mortality in severe traumatic brain injury with usage of β blocker

SECONDARY OUTCOMES:
Glascow outcome scale extended | 7 days
  Glascow outcome scale extended) consists of 8 categories:
  Death Persistent vegetative state: awake not aware. Lower severe disability: dependent, require help most of time. Upper severe disability: dependent, can be left alone some time. Iower moderate disability: independent, unable to work. Upper moderate disability: independent, reduced work capacity. Lower good recovery: minor problems that affect daily activities. Upper good recovery: no current problems related to brain injury.

CONTACTS AND LOCATIONS:
Overall Officials: Huda Elkallaf, Resident, Principal Investigator — Tanta University
Locations (1):
- Tanta University, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon reasonable request from principle investigator
Supporting Information: Study Protocol, SAP, ICF
Time Frame: For one year